CLINICAL TRIAL: NCT01641458
Title: Pharmacogenetics and Therapeutic Drug Monitoring for the Optimization of Fluoropyrimidine Treatment in Patients With Advanced Colorectal Cancer
Brief Title: Pharmacology-driven Dosing of Fluoropyrimidines in Cancer Patients
Acronym: FLOXTOX2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: University of Bern (Other)
Responsible Party: Principal Investigator, Markus Joerger, PD Dr. med. et phil II, Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG 343/12
Record Dates: First submitted 2012-07-11; First posted 2012-07-16 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Colorectal Cancer
Keywords: Genotyping; Area-under-the concentration-time curve; Toxicity; 5-fluorouracil; Capecitabine
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fluoropyrimidine-based chemotherapy (Experimental): DPYD-genotype and TDM-driven dosing of 5FU/Capecitabine
  Interventions: Other: 5FU and capecitabine (Xeloda®) dosing based on DPYD genotype; Other: Therapeutic drug monitoring of 5FU

INTERVENTIONS:
Other: 5FU and capecitabine (Xeloda®) dosing based on DPYD genotype — Multiplex amplification of each sample is performed in an individual well of a 24-well plate using a Mastercycler platform. Template and Platinum Taq Polymerase (Life Technologies, Carlsbad, California) are added to an analyte-specific amplification mix (AutoGenomics Inc., Carlsbad, California). After amplification, the plate is transferred into the Infinity analyzer (AutoGenomics Inc.), followed by primer extension and hybridization of detection primers to individual oligonucleotides arrayed on the Bio-FilmChip. After hybridization, the BioFilmChips are washed and scanned in the Infiniti optics module. The Autogenomics DPYD assay is used to detect the presence of the four risk alleles (IVS14+G>A, c.1679T>G, HapB3/c.1129-5923C>G and c.2846A>T).
Other: Therapeutic drug monitoring of 5FU — Repeated PK plasma sampling is done in all patients receiving 5FU. Blood is taken from venipuncture into one 5 ml heparin tube and into one 3 ml EDTA tube for the analysis of 5FU steady-state plasma concentrations in every (2-weekly) treatment cycle. Special attention has to be paid not to take PK blood from the site of drug infusion. For 5FU, PK sampling is done two hours before the calculated end of the 5FU pump on day 3 of every treatment cycle. The quantitative 5FU exposure expressed as the area-under-the concentration-time curve in mg•h/L is calculated from the measured steady-state plasma concentrations of 5FU and the duration of 5FU infusion. In all patients, 5FU doses for the second and subsequent administrations are adjusted to target a 5FU AUC between 20 and 30 mg•h/L

SUMMARY:
The fluoropyrimidines 5-fluorouracil (5FU) and capecitabine (Cp) are among the most commonly used anticancer drugs. Still, there is much controversy about the correct dosing, and the fact that a minority of patients experience severe, sometimes even lethal toxicity following treatment. One important factor predisposing patients to severe toxicity is deficiency in the 5FU-catabolic enzyme dihydropyrimidine dehydrogenase (DPD). Our group identified 4 DPD risk alleles in over 300 Swiss cancer patients, that resulted in a 8-times increased risk of experiencing severe toxicity from 5FU or Cp. In patients receiving 5FU as a continuous infusion, there are accumulating data that keeping the AUC of 5FU between 20-30 mg*h/L is beneficial in terms of treatment toxicity and activity. In this study, patients carrying at least 1/4 DPD risk alleles will receive a 50% dose reduction of either 5FU or Cp, with the potential of later dose increases in the abscence of severe toxicity. Additionally, patients receiving i.v. 5FU will undergo therapeutic drug monitoring at the end of the 2-day continuous infusion, with subsequent dose adaptations to target a 5FU AUC of 20-30 mg*h/L. The primary study objective is to reduce the incidence of severe treatment-related toxicity from 13% (in historical controls) to 5% in study patients.

ELIGIBILITY:
Inclusion Criteria:

* Cytological or histological proven diagnosis of colorectal cancer, metastatic or inoperable advanced disease, not amenable to curative therapy
* Measurable disease, defined as at least one lesion (outside of irradiated areas) that can be measured in at least one dimension as ≥ 10 mm (≥ 15 mm in case of lymph nodes) according to RECIST v1.1
* Tumor either wild-type KRAS or KRAS-mutated
* Indication for the therapeutic use of continuous intravenous 5FU over 48 hours ("deGramont" regimen) or oral Cp, either alone or in combination with other anticancer drugs (including monoclonal antibodies or other molecularly-targeted drugs)
* Eligible treatment regimens include: FOLFOX (FOLFOX 4, FOLFOX 6, modified FOLFOX 6, FOLFOX 7), FOLFIRI, 5FU or Cp mono-chemotherapy ("deGramont" regimen), XELOX, XELIRI, Capecitabine mono-chemotherapy
* All regimens may be combined with anti-VEGF or anti-EGFR targeted treatment such as bevacizumab or cetuximab
* Patients receive first-line systemic treatment (previous adjuvant chemotherapy is allowed, previous rectal radiochemotherapy is allowed if completed >/=1 months before registration to the study)
* Written informed consent before registration to the trial
* The patient is willing to undergo pharmacogenetic and pharmacokinetic sampling and analysis
* WHO performance status 0 or 1
* Female or male patients >18 years of age
* Adequate organ function (ANC, PLT, bilirubin 2xULN, creatinine clearance)

Exclusion Criteria:

* Known hypersensitivity to trial drug or any compounds of the drug
* Pregnant or breastfeeding women
* Patients with cerebral and/or leptomeningeal metastases are eligible, unless there is a need for treatment with steroids
* Risk of rapid deterioration due to tumor symptoms or tumor complications
* Severe or uncontrolled cardiovascular disease (e.g. ACS, cardiac failure NYHA III or IV, clinically relevant myopathy, history of myocardial infarction within the last 12 months, significant arrhythmias)
* Concurrent use of reversible or irreversible DPD-inhibitors, including brivudin, sorivudin, eniluracil 5-chloro-2,4-dihydroxypyridine or with substances interfering with the immunoassay, including theophylline and theobromine.
* Concurrent severe uncontrolled medical illness (judged by the investigator) which could impair the ability of the patient to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Predefined fluoropyrimidine-related (index) toxicity | After 6 weeks of fluoropyrimidine-based treatment
  Index toxicity is defined as follows:
  * All adverse events CTC grades ≥3, including myelosuppression but excluding nausea and vomiting (that is often due to concurrent platinum drug treatment)
  * Fluoropyrimidine-related toxicity CTC grade ≥2, including mucositis, dehydration, hand-foot syndrome
  * Diarrhea CTC grade ≥2 lasting for >/=5 days or an increase of 2 CTC grades in case of preexisting diarrhea. Diarrhea should not be evaluated in patients with a colostomy

SECONDARY OUTCOMES:
Area-under-the plasma-concentration time curve of 5-fluorouracil | at 8 weeks
  AUC of 5FU as derived from 5FU steady-state plasma concentrations, taken 2 hours before the planned end of the continuous drug infusion. 5FU target AUC is defined as within the range of 20-30 mg•h/L
Endogenous dihydrouracil/uracil ratio in plasma | at start of each treatment cycle
  Endogenous UH2 to U ratio as analysed at the time of PK sampling of 5FU or Cp, and repeated for each treatment cycle.
Objective treatment response (best response) according to RECIST v.1.1 | end of first-line treatment
  Objective treatment response according to the RECIST criteria v1.1 is assessed in all patients
Progression-free survival | time of disease progression or death
  Defined as the time interval between start of study treatment and disease progression or death, whatever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Joerger, MD PhD, Study Chair — Cantonal Hospital of St. Gallen
Locations (2):
- Switzerland (2):
  - Inselspital, Bern
  - Cantonal Hospital, Sankt Gallen